CLINICAL TRIAL: NCT03242096
Title: Treatment of Coronary In-stent Restenosis (ISR) by a Sirolimus Coated SEQUENT® SCB RAPID EXCHANGE PTCA Balloon Catheter or a Paclitaxel Coated SEQUENT® PLEASE PTCA Balloon Catheter
Brief Title: Treatment of Coronary In-stent Restenosis (ISR) by a Sirolimus Coated or a Paclitaxel Coated Balloon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InnoRa GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SI-ISR-01
Record Dates: First submitted 2017-07-31; First posted 2017-08-08 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Coronary Restenosis
MeSH Terms: conditions — Coronary Restenosis

STUDY DESIGN:
Intervention Model Description: Experimental intervention: Predilatation of coronary ISR with POBA followed by a sirolimus coated SeQuent® SCB balloon balloon (sirolimus 4.0 μg/mm²)
  Control intervention: Predilatation of coronary ISR with POBA followed by a paclitaxel coated SeQuent® Please balloon or SeQuent® Please NEO balloon (paclitaxel 3.0 μg/mm²)
Who Masked: Outcomes Assessor
Masking Description: Blinded QCA for primary outcome
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sirolimus coated balloon (Experimental): Treatment of in-stent restenosis with a sirolimus coated balloon
  Interventions: Combination Product: Sirolimus coated balloon
- Paclitaxel coated balloon (Active Comparator): Treatment of in-stent restenosis with a paclitaxel coated balloon
  Interventions: Combination Product: Paclitaxel coated balloon

INTERVENTIONS:
Combination Product: Sirolimus coated balloon — Predilatation of coronary ISR with POBA (balloon-to-stent ratio 1:1) followed by a sirolimus coated balloon (SeQuent®SCB balloon with sirolimus 4.0 μg/mm²)
  Arms: Sirolimus coated balloon
Combination Product: Paclitaxel coated balloon — Predilatation of coronary ISR with POBA (balloon-to-stent ratio 1:1) followed by a paclitaxel coated balloon (SeQuent®Please balloon or SeQuent®Please NEO balloon with paclitaxel 3.0 μg/mm²) (paclitaxel 3.0 μg/mm²)
  Arms: Paclitaxel coated balloon

SUMMARY:
Treatment of coronary in-stent restenosis (ISR) by a sirolimus coated SEQUENT® SCB RAPID EXCHANGE PTCA balloon catheter or a paclitaxel coated SEQUENT® PLEASE PTCA balloon catheter

DETAILED DESCRIPTION:
Experimental intervention: Predilatation of coronary ISR with POBA followed by a sirolimus coated SeQuent®SCB balloon balloon (sirolimus 4.0 μg/mm²)

Control intervention: Predilatation of coronary ISR with POBA followed by a paclitaxel coated SeQuent®Please balloon or SeQuent®Please NEO balloon (paclitaxel 3.0 μg/mm²)

Duration of intervention per patient: minutes

Follow-up per patient: 30 days telephone call; 6 months angiographic + 12 months clinical follow up

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Clinical evidence of stable or unstable angina (acute coronary syndrome) or a positive functional study
* Patients with ≤ 2 primary in-stent restenosis (ISR) lesions (≥ 70% diameter stenosis by visual estimation or ≥50% and positive functional study) including margin-stenosis with max 5 mm distance to the stent

Exclusion Criteria:

* Chronic renal insufficiency with serum creatinine levels > 2.0 mg per deciliter
* Known hypersensitivity or contraindications to aspirin, heparin, clopidogrel, ticlopidine or sirolimus, and sensitivity to contrast media not amenable to premedication
* Concomitant medical illness associated with a life-expectancy of less than two year
* Lesion length (ISR) > 35 mm, reference vessel diameter < 2.5 mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
late lumen loss in-lesion at 6 months | 6 months
  late lumen loss in-lesion at 6 months assessed by blinded QCA

SECONDARY OUTCOMES:
Procedural Success | during hospital stay of index procedure
  < 30% final stenosis, TIMI III flow, no flow-limiting dissection, and the absence of in-hospital MACE
MACE | 6 and 12 months
  cardiac death, target vessel myocardial infarction, and clinically driven target lesion revascularization
Individual clinical endpoints | 6 and 12 months
  stent thrombosis, cardiac death, target lesion myocardial infarction, clinically driven target lesion revascularization, binary restenosis (stenosis ≥ 50% at follow-up angiography)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Scheller, MD, Principal Investigator — University of Saarland
Locations (5):
- Germany (4):
  - Clinical and Experimental Interventional Cardiology, Homburg, Saarland
  - Klinik für Innere Medizin und Kardiologie, Dresden
  - Deutsches Zentrum für Herz und Kreislauf, Mainz
  - Dept. of Internal Medicine II, Ulm
- Universitätsspital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Scheller B, Hehrlein C, Bocksch W, Rutsch W, Haghi D, Dietz U, Bohm M, Speck U. Treatment of coronary in-stent restenosis with a paclitaxel-coated balloon catheter. N Engl J Med. 2006 Nov 16;355(20):2113-24. doi: 10.1056/NEJMoa061254. Epub 2006 Nov 13. PMID 17101615
- [Derived] Scheller B, Mangner N, Abdul Kader MASK, Wan Ahmad WA, Jeger R, Wohrle J, Ong TK, Liew HB, Gori T, Mahfoud F, Nuruddin AA, Woitek F, Abidin IZ, Schwenke C, Schnorr B, Mohd Ali R. Combined Analysis of Two Parallel Randomized Trials of Sirolimus-Coated and Paclitaxel-Coated Balloons in Coronary In-Stent Restenosis Lesions. Circ Cardiovasc Interv. 2022 Sep;15(9):e012305. doi: 10.1161/CIRCINTERVENTIONS.122.012305. Epub 2022 Sep 20. PMID 36126132